CLINICAL TRIAL: NCT06440616
Title: Benefit of Spectral Information Provided by Photon Counting CT in Patients Suspected for Lung Cancer
Brief Title: Benefit of Spectral Information in Patients Suspected for Lung Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Copenhagen University Hospital at Herlev (Other)
Collaborators: Rigshospitalet, Denmark (Other); Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Michael Brun Andersen, Associate Professor, PhD, Copenhagen University Hospital at Herlev
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: H- 23045674
Record Dates: First submitted 2024-05-27; First posted 2024-06-04 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Lung Neoplasm Malignant
Keywords: Computed tomography; Spectral CT
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CT images without spectral information available (No Intervention): Reported without access to spectral information in a normal clinical practice. Supplemental examinations suggested as per the ACR white papers for incidental findings.
- CT images with spectral information available (Experimental): Reported with access to spectral information in a normal clinical practice. Supplemental examinations suggested as per the ACR white papers for incidental findings.
  Interventions: Device: Spectral CT images generated by a photon counting CT scanner

INTERVENTIONS:
Device: Spectral CT images generated by a photon counting CT scanner — The reading radiologist will in the experimental arm have access to spectral CT images in the form of low virtual monoenergetic images, virtual non-contrast images, iodine maps and effective atomic number. In the non-interventional arms the reading radiologist will only have access to conventional CT images.
  Arms: CT images with spectral information available

SUMMARY:
Purpose The aim of the study is to investigate the utilization of photon counting CT (PCCT) and the spectral information provided to determine the impact of spectral information on follow-up examinations.

As secondary aims we will compare conventional CT, CT + 18Flouro-deoxy-glucose (18F-FDG) positron emission tomography (PET) and PCCT + 18F-FDG PET for the tumor-node-metastasis (TNM) staging of lung cancer patients.

PCCT with and without spectral information to assess the need for additional work-up,TNM classification, and sensitivity/specificity for malignant lesions. Patients will be randomized for reading with or without spectral information available within a clinical setting. The clinical readings are performed as a structured reports of all significant findings. Including both malignant and benign findings. Furthermore, in case additional follow-up/work-up is needed based on the guidelines on incidental findings by the American College of Radiology (ACR), this will be reported as well. If lesions suspicious of pulmonary malignancy is present, a provisional TNM classification is provided based on the scan findings.

After 3 months, the patient record is reviewed where additional examinations that can be attributed to the PCCT scan are recorded. The financial impact is calculated by a health economist based on the findings. PET/CT, conventional CT and PCCT combined with PET will be assessed retrospectively for comparison. Endpoints are number of supplementary examinations and cost savings. Sensitivity and specificity for any malignant finding. The T, N and M stages are assessed separately as diagnostic measures by the McNemar's test with a reference standard from the Danish Lung cancer register. The number of malignant lesions will be determined by reviewing the patient records incl. pathology assessment if available 12 months after inclusion of the last patient.

ELIGIBILITY:
Inclusion Criteria:

* Patients suspected of lung cancer refered to Copenhagen University Hospital as per the guidelines from the danish national health authorities from either the general practitioner or from the department of pulmonology.
* Informed consent

Exclusion Criteria:

* Patients who cannot tolerate intravenous iodinated contrast
* Already verified lung cancer from another institution
* Comorbidities that exclude the patient from receiving treatment
* Lack of reference standard in the form of either histology or follow-up
* Known extrapulmonary malignancy
* Technical limitations within the scans/reconstructions
* other

Pr. the 29th of September included 433 participants.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2024-05-24 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Number of follow up examinations | Baseline
  Determine the number of suggested follow-up examinations based on the initial CT scan to learn the significance of spectral information in a clinical setting.

SECONDARY OUTCOMES:
T, N, and M stage | 24 months
  Determine the accuracy of T, N, and M stage based on PCCT, conventional CT, PET/CT and PET/PCCT. Retrospective assessment 24 months after primary scan.
Number of malignant lesions | 24 months
  Determine the number of found malignant lesions in each arm. Reference standard will be follow up or pathology within a minimum of one year of the scan. That means 12 months after the end of the inclusion period.

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Andersen, PhD, Principal Investigator — Copenhagen University Hospital at Herlev
Locations (1):
- Copenhagen University Hospital Herlev, Herlev, Capital Region, Denmark

IPD SHARING:
Plan to Share IPD: No